CLINICAL TRIAL: NCT03169998
Title: The Effect of Goal-directed Fluid Therapy on Postoperative Complications in Patients Undergoing Laparoscopic Hepatobiliary or Pancreatic Surgery
Brief Title: Effect of Goal-directed Fluid Therapy on Postoperative Complications
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Clinical professor, Seoul National University Bundang Hospital
Other Study IDs: EV1000
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Liver Diseases; Pancreas Disease
MeSH Terms: conditions — Liver Diseases; Pancreatic Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GDFT group: The fluid infusion is to be performed, in accordance with GDFT protocol, on the basis of cardiac index (CI), stroke volume index(SVI) and stroke volume (SV) in addition to invasively measured arterial pressure by Vigilio / FloTrac Monitor.
  Interventions: Device: EV1000 platform
- Control group: Patients in whom the surgery was conducted without the use of EV1000/ FloTrac monitoring among those who had undergone laparoscopic hepatobiliary or pancreatic surgery in the past.

INTERVENTIONS:
Device: EV1000 platform — a continuous arterial pressure monitoring was performed via EV1000/ FloTrac (Edwards Lifesciences, Irvine, CA, USA) (Fig 1) with the continuous monitoring of cardiac index (CI), stroke volume index (SVI) and stroke volume (SV).
  Groups: GDFT group

SUMMARY:
* It has been known that the recent application of a goal-directed fluid therapy (GDFT) to the intraoperative fluid infusion in patients contributes to decreasing the prevalence of postoperative complications and shortening the length of study in the intensive care unit as well as hospital stay compared with conventional methods.
* Laparoscopic surgery is in a trend that its application is being expanded recently, but there has been no report on the application of GDFT to laparoscopic surgery so far.
* To this end, this study aims to apply the intraoperative GDFT protocol in patients undergoing laparoscopic hepatobiliary or pancreatic surgery and to find out whether there is any difference in postoperative recovery and incidences of postoperative complications, by comparing with patients applied with the fluid therapy using existing conventional methods

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic hepatobiliary or pancreatic surgery

Exclusion Criteria:

* Patients who do not consent to participation in the study
* Pregnant women, breastfeeding women

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is to be conducted in patients scheduled with laparoscopic hepatobiliary or pancreatic surgery, who are at risk either for taking 2 hours or more in surgery or to lose blood of 1000 ml or more.
Sampling Method: Non-Probability Sample
Enrollment: 375 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Pulmonary complication | Postoperative 90 day
Wound complication | Postoperative 90 day
Acute kidney injury | Postoperative 90 day
Delirium | Postoperative 90 day
Deep vein thrombosis | Postoperative 90 day
Myocardiac infarction | Postoperative 90 day
Stroke | Postoperative 90 day
Sepsis | Postoperative 90 day
Urinary tract infection | Postoperative 90 day
Death | Postoperative 90 day

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea